CLINICAL TRIAL: NCT05284539
Title: Efficacy of Platinum-based Chemotherapy With or Without Immune Checkpoint Inhibitors in Patients With EGFR/ALK/ROS1 Sensitive Mutated NSCLC Who Progressed From Previous Tyrosine Kinase Inhibitors (TKI) Therapy
Brief Title: Efficacy of Platinum-based Chemotherapy Plus Immune Checkpoint Inhibitors for EGFR/ALK/ROS1 Mutant Lung Cancer
Acronym: Awesome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Head of Medical Oncology, Director of Early Clinical Trial Center, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220117
Record Dates: First submitted 2022-01-22; First posted 2022-03-17 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: EGFR; ALK; ROS1; PD-1 Blockade
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Bevacizumab; pembrolizumab; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: EGFR mutant Group (Experimental): EGFR mutant Group.
  Interventions: Drug: Pemetrexed, Cisplatin, Bevacizumab Plus Pembrolizumab
- Arm B: ALK fusion Group (Experimental): ALK fusion Group.
  Interventions: Drug: Pemetrexed, Cisplatin, Bevacizumab Plus Pembrolizumab
- Cohort C: ROS1 fusion Group. (Experimental): ROS1 fusion Group.
  Interventions: Drug: Pemetrexed, Cisplatin, Bevacizumab Plus Pembrolizumab

INTERVENTIONS:
Drug: Pemetrexed, Cisplatin, Bevacizumab Plus Pembrolizumab — Pemetrexed, 500mg/m2, ivgtt, every 21 days. Bevacizumab 15mg/kg, ivgtt, every 21 days. Pembrolizumab, 200mg ivgtt, every 21 days. Atezolizumab, 1200mg, ivgtt, every 21 days.
  Other Names: Pemetrexed; Bevacizumab; Pembrolizumab; Atezolizumab

SUMMARY:
The investigators want to evaluate the Efficay and Safety of Platinum-based Chemotherapy with or without immune checkpoint inhibitors for EGFR/ALK/ROS1 Positive NSCLC who Failed from First-Line Standard Treatment.

DETAILED DESCRIPTION:
The investigators want to evaluate the Efficacy and Safety of Platinum-based Chemotherapy with or without immune checkpoint inhibitors for EGFR/ALK/ROS1 Positive NSCLC who Failed from First-Line Standard Treatment.

This study will be divided into three cohorts. Cohort A for EGFR mutation NSCLC, Patient with NGS identified EGFR sensitive mutation NSCLC who failed from first line Osimertinib will be included.

Cohort B for ALK fusion NSCLC, Patient with NGS identified ALK fusion NSCLC who failed from first line Alectinib/Lorlatinib/Ceritinib/Ensartinib/Brigatinib will be included. All the patients will be divided two group,3'ALK and 3'ALK with retention of 5'ALK.

Cohort C for ROS1 fusion NSCLC, Patient with NGS identified ROS1 fusion NSCLC who failed from first line Crizotinib/Entrectinib/Ensartinib/Brigatinib will be included.

The investigators will collect the safety and efficacy data for all the patients.

The tissue and blood samples will be collected under the permission of the participate.

Single cell sequencing, DSP, RNA-seq and IHC will be performed to evaluate the TME.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the requirements and contents of the clinical trial, and provide a signed and dated informed consent form.
2. Age ≥ 18 years.
3. Histologically or cytologically confirmed, Stage IV NSCLC.
4. EGFR/ALK/ROS1-sensitive mutations confirmed by an accredited local laboratory, progressed from first line systematic therapy.
5. ECOG 0-1.
6. Predicted survival ≥ 12 weeks.
7. Adequate bone marrow hematopoiesis and organ function
8. Presence of measurable lesions according to RECIST 1.1.

Exclusion Criteria:

Cancer-Specific Exclusions:

* Active or untreated central nervous system metastases.
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome.

General Medical Exclusions:

* Pregnant or lactating women.
* History of autoimmune disease.
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Positive test for human immunodeficiency virus.
* Active hepatitis B or hepatitis C.
* Severe infection within 4 weeks prior to randomization.
* Significant cardiovascular disease.
* Illness or condition that interferes with the participant's capacity to understand, follow and/or comply with study procedures.

Exclusion Criteria Related to Medications:

• Prior treatment with cluster of differentiation 137 agonists or immune checkpoint blockade therapies, anti-programmed death-1, and anti-PD-L1 therapeutic antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from first subject dose to study completion, or up to 36 month
  To assess progression-free survival of patients treated with Immune Checkpoint Inhibitor, Bevacizumab in combination with Chemotherapy according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as first dose to first documented disease progression assessed by investigator or death due to any cause

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Time from first dose to last dose, or up to 24 month
  To assess PD-1 antibody, Bevacizumab in combination with Chemotherapy overall response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as the proportion of subjects who have a complete response (CR) or a partial response (PR)
Overall survival (OS) | Time from first subject dose to study completion, or up to 36 month
  To assess overall survival, define as first dose to the death of the subject due to any cause
Adverse events (AEs) according to CTCAE 5.0 | From first dose until 28 days after the last dose, up to 24 month
  Number of participants with adverse events (AEs) according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China